CLINICAL TRIAL: NCT04230200
Title: A Large-scale, Prospective Screening Programme for Malignant Tumors Using Routine Blood Tests Parameters
Brief Title: Prospective Screening Programme for Malignant Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, President, Sun Yat-sen University
Other Study IDs: SCREEN-Pan Cancer
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Hematologic Tests; Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy cohort: People who received routine physical examination including blood test, and after 3 year follow-up, have not been diagnosed as any kind of malignant tumor.
- Malignancy Cohort: People who were diagnosed as one of the following malignant disease: breast cancer, lung cancer, gastric cancer， esophageal cancer，colorectal cancer，nasopharyngeal cancer，liver cancer and cervical cancer

SUMMARY:
In prospective part of study, the investigators have found that the parameters of routine blood tests can differentiate varieties of malignancy from healthy people.

The investigators enrolled healthy subjects and patients with malignancy that aged from 18 to 85，and collected their clinical data and blood tests result to build the model.And retrospectlly enroll healthy subjects and patients to test the model.

ELIGIBILITY:
For the cohort of healthy people

Inclusion Criteria:

1. Asymptomatic persons between the ages of 18 to 80 years
2. Chinese ethnicity
3. After 3 year follow-up, diagnosed with no malignant disease
4. Subject underwent routine blood tests in our center

Exclusion Criteria:

1.With a history of malignant disease

For the cohort of patients with malignancy

Inclusion Criteria:

1. diagnosis with the following malignant disease，breast cancer, lung cancer, gastric cancer， esophageal cancer，colorectal cancer，nasopharyngeal cancer，liver cancer and cervical cancer
2. Subject underwent routine blood tests in our center

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Malignant tumor is a common Threat to human health worldwide. Some of the routine blood tests parameters were reportedly predictive of the risk of Malignant tumor. This study aims to investigate whether routine blood tests parameters would be useful in the screening of Malignant tumor in asymptomatic individuals.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity (true positive rate) | 1 year
  The proportion of persons with disease who have a positive test (positive test results among persons with disease)
Specificity (true negative rate) | 1 year
  The proportion of persons without disease who have a negative test (negative test results among persons without disease)

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Heimbach JK, Kulik LM, Finn RS, Sirlin CB, Abecassis MM, Roberts LR, Zhu AX, Murad MH, Marrero JA. AASLD guidelines for the treatment of hepatocellular carcinoma. Hepatology. 2018 Jan;67(1):358-380. doi: 10.1002/hep.29086. No abstract available. PMID 28130846
- [Background] Chan KCA, Woo JKS, King A, Zee BCY, Lam WKJ, Chan SL, Chu SWI, Mak C, Tse IOL, Leung SYM, Chan G, Hui EP, Ma BBY, Chiu RWK, Leung SF, van Hasselt AC, Chan ATC, Lo YMD. Analysis of Plasma Epstein-Barr Virus DNA to Screen for Nasopharyngeal Cancer. N Engl J Med. 2017 Aug 10;377(6):513-522. doi: 10.1056/NEJMoa1701717. PMID 28792880